CLINICAL TRIAL: NCT02950935
Title: Prospective, Double-blind, Randomised, Placebo Controlled, Phase III Clinical Study Assessing the Efficacy of Natural Progesterone 25 mg/Bid Administered Subcutaneously in the Maintenance of Early Pregnancy in Women With Symptoms of Threatened Abortion
Brief Title: Progesterone in Threatened Abortion
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16I-Prg06
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Threatened Abortion in First Trimester
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progesterone (Experimental): 25 mg of subcutaneous progesterone will be administered twice à day until the 12th week of gestation.
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): placebo will be administered twice à day until the 12th week of gestation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — subcutaneous injection of progesterone solution will be performed twice à day from onset of threatened abortion symptoms until week 12 of pregnancy.
  Arms: Progesterone
Drug: Placebo — subcutaneous injection of placebo solution will be performed twice à day from onset of threatened abortion symptoms until week 12 of pregnancy.
  Arms: Placebo

SUMMARY:
The main objective of this study will be to assess the efficacy of natural progesterone at a daily dose of 25 mg/bid in the maintenance of early pregnancy in women with symptoms of threatened abortion. The secondary objectives will be the efficacy of progesterone in reducing both pain and uterine contractions.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending the emergency room of the study sites with the following characteristics:
* Able and willing to sign the Subject Informed Consent Form and adhere to the study visit schedule;
* Age: 18-37 years;
* BMI: 18-28 kg/m2;
* Symptoms of threatened abortion (vaginal bleeding , with or without pelvic pain);
* Ultrasound proof of viable singleton intrauterine pregnancy (positive foetal heart beat);
* Gestation week ≥6 weeks (5 w +1d) and <12 weeks (11 w + 1d) according to ultrasound dating (CRL);
* Closed uterine cervix;
* At the first case of threatened abortion in the current pregnancy.

Exclusion Criteria:

* Pregnancy obtained via ART treatment;
* Subchorionic haematoma with >50% placental detachment;
* History of recurrent miscarriage;
* Severe uterine malformations;
* Known hypersensitivity to study medication;
* Neoplasias (known or suspected breast or genital tract cancer);
* Severe impairment of hepatic or renal function;
* Use of concomitant medications that might interfere with study evaluations (other hormonal treatment or drugs affecting uterine contractility);
* Active arterial or venous thromboembolism or severe thrombophlebitis, or a history of these events;
* Porphyria;
* A history of idiopathic jaundice, severe pruritus or pemphigoid gestationis during pregnancy;
* Antiphospholipid syndrome;
* Diabetes mellitus;
* Known thyroid diseases or autoimmune conditions.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate at 12 weeks of gestation | 12 weeks

SECONDARY OUTCOMES:
Reduction of the frequency of uterine contractions; | 15 days
Pain reduction (using a Numerical Rating Scale); | 15 days
Reduction of subchorionic haematoma; | 15 days
  Size of subchorionic haematoma will be measured (in mm) at screening and after treatment.
Number of subjects with onset of new threatened abortion | 12 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - "F. Miulli" Regional General Hospital, Bari, BA
  - P.O.G. Salesi, Ancona
  - Ospedale Cervesi, Cattolica
  - Presidio Ospedale S'Anna, Torino